CLINICAL TRIAL: NCT03047772
Title: The Randomized Double-blind Placebo-Controlled Multi-center Clinical Trial of Transplantation Efficacy of Autologous Bone Marrow Mesenchymal Stem Cells With Intensive Atorvastatin in Acute Myocardial Infarction Patients
Brief Title: Transplantation Efficacy of Autologous Bone Marrow Mesenchymal Stem Cells With Intensive Atorvastatin in AMI Patients
Acronym: TEAM-AMI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuejin Yang (Other)
Collaborators: Peking Union Medical College Hospital (Other); The First Hospital of Hebei Medical University (Other); Zunyi Medical College (Other)
Responsible Party: Sponsor-Investigator, Yuejin Yang, Vice Dean of Fuwai hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-807-10.1
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Infarction; Stem Cell Transplantation; Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: conditions — Myocardial Infarction | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase A: Atorvastatin (Placebo Comparator): Atorvastatin routine dose + placebo transplantation
  Interventions: Drug: Atorvastatin
- Phase A: Low dose BMMSC (Experimental): Atorvastatin routine dose + low dose BMMSC Transplantation
  Interventions: Drug: Atorvastatin; Drug: Low dose BMMSC
- Phase A: Middle dose BMMSC (Experimental): Atorvastatin routine dose + middle dose BMMSC Transplantation
  Interventions: Drug: Atorvastatin; Drug: Middle dose BMMSC
- Phase A: High dose BMMSC (Experimental): Atorvastatin routine dose + high dose BMMSC Transplantation
  Interventions: Drug: Atorvastatin; Drug: High dose BMMSC
- Phase B: Atorvastatin (Placebo Comparator): Atorvastatin routine dose + placebo transplantation
  Interventions: Drug: Atorvastatin
- Phase B: Atorvastatin+Transplantation (Active Comparator): Atorvastatin routine dose+ Optimal dose BMMSC Transplantation
  Interventions: Drug: Atorvastatin; Drug: Transplantation
- Phase B: Intensive Atorvastatin (Placebo Comparator): Atorvastatin Intensive dose + placebo transplantation
  Interventions: Drug: Intensive Atorvastatin
- Phase B: Intensive Atorvastatin+Transplantation (Experimental): Atorvastatin Intensive dose + Optimal dose BMMSC Transplantation
  Interventions: Drug: Intensive Atorvastatin; Drug: Transplantation

INTERVENTIONS:
Drug: Atorvastatin — Routine dose of Atorvastatin therapy
  Other Names: Statin
  Arms: Phase A: Atorvastatin; Phase A: High dose BMMSC; Phase A: Low dose BMMSC; Phase A: Middle dose BMMSC; Phase B: Atorvastatin; Phase B: Atorvastatin+Transplantation
Drug: Intensive Atorvastatin — Intensive dose of Atorvastatin therapy
  Arms: Phase B: Intensive Atorvastatin; Phase B: Intensive Atorvastatin+Transplantation
Drug: Low dose BMMSC — Low dose autologous Bone Marrow Mesenchymal Stem Cells transplantation
  Arms: Phase A: Low dose BMMSC
Drug: Middle dose BMMSC — Middle dose autologous Bone Marrow Mesenchymal Stem Cells transplantation
  Arms: Phase A: Middle dose BMMSC
Drug: High dose BMMSC — High dose autologous Bone Marrow Mesenchymal Stem Cells transplantation
  Arms: Phase A: High dose BMMSC
Drug: Transplantation — Optimal dose autologous Bone Marrow Mesenchymal Stem Cells transplantation
  Arms: Phase B: Atorvastatin+Transplantation; Phase B: Intensive Atorvastatin+Transplantation

SUMMARY:
The benefit of current stem cell transplantation therapy for myocardial infarction is limited by low survival rate for stem cell. The purpose of this study is to test whether intensive Atorvastatin therapy can improve the outcome of patients with impaired left ventricle function after acute myocardial infarction who underwent intracoronary transfer of autologous bone marrow mesenchymal stem cells.

DETAILED DESCRIPTION:
The major challenge to a successful stem cell therapy for myocardial infarction is the low survival rate of implanted cells in the damaged tissue. Atorvastatin, an HMG-CoA reductase inhibitor, has multiple biological activities independent of cholesterol-lowering action.This study is performed to find out more information about the strategy with Atorvastatin therapy to improve the survival of implanted cells, autologous bone marrow mesenchymal stem cells transplantation. Patients between 30 and 75 years of age who receive autologous bone marrow mesenchymal stem cells transplant may be eligible for this study. These patients receive autologous bone marrow mesenchymal stem cells transplantation intracoronary undergoing Percutaneous Coronary Intervention with regular or high dose of Atorvastatin treatment. The objective evaluations will be performed at baseline and during 12 months follow-up.

Heart function tests may include the following:

Electrocardiogram (EKG) evaluates the electrical activity of the heart. Electrodes placed on the chest transmit information from the heart to a machine.

Echocardiogram (Echo) is an ultrasound test that uses sound waves to create an image of the heart and examine the function of the heart chambers and valves.

Gated acquisition scan is a nuclear medicine test that uses a small amount of radioactive chemical injected into a vein. A special scanner creates an image of the heart for examining the beating motion of the muscle.

MRI evaluates function of the heart chambers the beating motion of the muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the first time ST-elevation myocardial infarction (STEMI).
2. Patients after undergoing PCI 2 to 5 days.
3. Patients without PCI but emergency coronary angiography shows the criminal coronary artery recanalized.
4. Left ventricular infarction area seriously hypokinesis or no movement
5. Left ventricular ejection fraction <=45% based on coronary angiography or echocardiography.

Exclusion Criteria:

Any one of the following exclusion criteria is sufficient to disqualify a patient from the study.

1. Patients without emergency PCI and the criminal coronary artery fail to be recanalized.
2. Patients with non-ST-elevation myocardial infarction.
3. Patients with normal left ventricular function.
4. Patients with mechanical complications of myocardial infarction.
5. Patients with a malignant tumor.
6. Patients with infection disease.
7. Less than 6 months since last episode of stroke.
8. Patients with hematological disease (leukemia, myeloproliferative disease, or myelodysplastic syndromes).
9. ALT (GPT) exceeding 100 IU/L.
10. Leukocytes less than 4,000/µL or exceeding 10,000/µL.
11. Platelets less than 100,000/µL.
12. Hemoglobin less than 10 g/dL.
13. Pregnant or nursing patients, those who may be pregnant, or those who plan on becoming pregnant before the end of the study period.
14. Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-03-06 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction from baseline to 12 months' | 12 months
  Changes in left ventricular ejection fraction from baseline to 12 months' by MRI

REFERENCES:
- [Derived] Xu JY, Qian HY, Huang PS, Xu J, Xiong YY, Jiang WY, Xu Y, Leng WX, Li XD, Chen GH, Tang RJ, Huang CR, Hu MJ, Jin C, Wu Y, Zhang J, Qian J, Xu B, Zhao SH, Lu MJ, Shen R, Fang W, Wu WC, Chen X, Wang Y, Li W, Lu XF, Jiang XF, Ma CC, Li JW, Geng YJ, Qiao SB, Gao RL, Yang YJ. Transplantation efficacy of autologous bone marrow mesenchymal stem cells combined with atorvastatin for acute myocardial infarction (TEAM-AMI): rationale and design of a randomized, double-blind, placebo-controlled, multi-center, Phase II TEAM-AMI trial. Regen Med. 2019 Dec;14(12):1077-1087. doi: 10.2217/rme-2019-0024. Epub 2019 Dec 12. PMID 31829095